CLINICAL TRIAL: NCT04858139
Title: "Exploration de l'Effet Sur le métabolisme cérébral de l'Administration de Lactate après Accident Vasculaire cérébral Chez l'Homme" (French Title)
Brief Title: Exploring the Effect of Lactate Administration After Ischemic Stroke on Brain Metabolism
Acronym: LacAVC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment slow. Standard stroke patient management was changed (CT replacing MRI if NIHSS > 10). We closed the study to avoid bias (after 28 inclusions /out of 30 planned)
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Lorenz Hirt, MD, MD, associate professor, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Swissmedic N°2020DR2163; 2019-00897 (Other: CER-VD)
Record Dates: First submitted 2021-03-30; First posted 2021-04-26 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Lactic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Numbered vials, prepared by hospital pharmacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): patients will be injected with placebo
  Interventions: Drug: Placebo
- Lactate (Active Comparator): patients will be injected with lactate solution
  Interventions: Drug: Lactate

INTERVENTIONS:
Drug: Lactate — Intravenous injection (20 min), 300 mmol/L, 1mmol/Kg body weight,
  Arms: Lactate
Drug: Placebo — Intravenous injection (20 min)
  Other Names: Saline solution administration
  Arms: placebo

SUMMARY:
In this exploratory randomized double blind placebo controled trial, lactate solution or placebo will be administered to acute ischemic stroke patients selected for endovascular treatment (EVT) without intravenous thrombolysis. The treatment will be administered within one hour after EVT. Primary outcome measures will be lactate and metabolite concentrations in the ischemic lesion, in the penumbra and contralaterally, evaluated by magnetic resonance spectroscopy(MRS). Secondary outcome measures will be evolution of the ischemic penumbra, clinical outcome at 3 months.The trial will end when 10 patients per group have completed the study.

DETAILED DESCRIPTION:
This is an exploratory randomized double blind placebo controled trial on acute ischemic stroke patients. Lactate solution or placebo will be administered to acute ischemic stroke patients selected for endovascular treatment (EVT) without intravenous thrombolysis. Magnetic resonance spectroscopy will be performed before EVT to measure metabolite concentrations in the ischemic core, penumbra and in the contralateral hemisphere. The treatment will be administered within one hour after EVT. As soon as the patient is stabilized, she/he will undergo an additional magnetic resonance imaging (MRI) with magnetic resonance spectroscopy (MRS). MRS will also be performed during the control MRI after 24 hours. Neurological deficits will be evaluated on admission, at 24 hours using the National Institute of Health Stroke Scale (NIHSS), and at 3 months, with both NIHSS and the modified Rankin scale. Primary outcome measures will be lactate and metabolite concentrations changes in the ischemic lesion, in the penumbra and the contralateral side, evaluated by magnetic resonance spectroscopy after intervention compared to baseline MRS values. Secondary outcome measures will be evolution of the ischemic penumbra and clinical outcome at 3 months. The trial will end when 10 patients per group have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke with arterial occlusion affecting middle cerebral artery (segment M1or segment 2) or internal carotid artery (T-type or L-type occlusion) selected for EVT
* not eligible for intravenous thrombolysis (IVT)
* Moderate to severe stroke (NIHSS > or = 4), and preadmission mRS > or = 3)
* Perfusion - diffusion mismatch
* Obtain consent from independent Doctor Randomisation criteria
* If possible oral consent from patient or relatives
* Treatment administration possible within 1h from EVT

Exclusion Criteria:

* Rapid neurological recovery
* Clinically unstable patient
* Contraindications to MRI
* Blood Na+ > 155 mmol/l or plasma osmolality > 320 mosmol/l
* Medical history of traumatic brain injury (TBI), neurodegenerative disease, intracranial hemorrhage, cerebral aneurysm, brain tumour
* Medical history of psychiatric disorders
* Liver insufficiency
* Heart failure
* Pregnancy (pregnancy test required in women aged under 50 unless patient or relatives indicate that the patient is not pregnant)
* Participation in another clinical trial in the last 30 days
* Lack of consent of an independent Doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Does the administered lactate reach the brain | Measurement after intervention (as soon as the patient condition allows performing an MRI; estimated between 1 and 2 hours)
  Measurement of lactate and other metabolites in lesion, penumbra, contralateral side using magnetic resonance spectroscopy measured after intervention and compared to baseline values.
  After intervention, the MRS will be performed as soon as possible considering that these patients have an EVT under general anesthesia and need to be stabilised after the EVT and study treatment intervention before the MRS.
Does the administered lactate persist in the brain at 24 hours | The MRS will be performed during the routine clinical MRI approximately 24 hours after EVT
  Measurement of lactate and other metabolites in lesion, penumbra, contralateral side using magnetic resonance spectroscopy measured at 24 hours and compared to baseline values.

SECONDARY OUTCOMES:
Effect of lactate on neuronal death after intervention | Measurement after intervention (as soon as the patient condition allows performing an MRI; estimated between 1 and 2 hours)
  Assessment of N-acetyl aspartate (NAA), a neuronal marker, using MRS and compared to baseline values, in the ischemic core and in the ischemic penumbra.
Effect of lactate on neuronal death at 24 hours | Measurement at during the routine control MRS, approximately 24 hours after EVT
  Assessment of N-acetyl aspartate (NAA), a neuronal marker, using MRS and compared to baseline values, in the ischemic core and in the ischemic penumbra.
Effect of lactate on evolution of lesion at 24 hours | At 24 hours
  Assessment of lesion using diffusion weighted Imaging (DWI) compared to baseline value
Effect of lactate on evolution of penumbra at 24 hours | This evaluation will be based on the routine MRI evaluation performed approximately 24 hours after EVT
  Check impact of intervention on the penumbra using perfusion weighted imaging (PWI) at 24 hours compared to baseline
Clinical outcome at 24 hours | at 24 hours
  Evolution of the neurological score (NIHSS) and compared to baseline assessment
Clinical outcome at 3 months | Measurement at follow up (3 months)
  Evolution of neurological score (NIHSS) compared to baseline value
Handicap at 3 months | Measurement at follow up (3 months)
  Evolution of neurological handicap (mRS) compared to baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Hirt, MD, Principal Investigator — CHUV
Locations (1):
- CHUVaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual patient data will be made available 1 year after the end of the study to other investigators if the patient provides informed consent for further use of his/her data.